CLINICAL TRIAL: NCT03477006
Title: Pragmatic Prehospital Group O Whole Blood Early Resuscitation (PPOWER) Trial: A Prospective, Interventional,Randomized, 3 Year, Pilot Clinical Trial
Brief Title: Pragmatic Prehospital Group O Whole Blood Early Resuscitation Trial
Acronym: PPOWER
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow enrollment, financial considerations and global pandemic
Sponsor: Jason Sperry (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Jason Sperry, Professor of Surgery and Critical Care Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34HL135224 (NIH); R34HL135224 (NIH)
Record Dates: First submitted 2018-03-19; First posted 2018-03-26 (Actual); Results first posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Hemorrhagic Shock
MeSH Terms: conditions — Shock, Hemorrhagic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LTLR-WB (Experimental): Receiving 2 units of low titer, leucocyte reduced, platelet replete whole blood initiated in the prehospital setting during air medical transport and continued (up to 6 units of whole blood followed by standard component resuscitation) thru the early in-hospital phase of care
  Interventions: Biological: Whole blood
- Standard Care (No Intervention): Receiving standard prehospital air medical care and standard of care component (1:1:1) trauma resuscitation thru the early in-hospital phase of care

INTERVENTIONS:
Biological: Whole blood — Low titer, group O, leukocyte reduced, platelet replete, cold stored whole blood
  Arms: LTLR-WB

SUMMARY:
Despite advances in trauma resuscitation, a paucity of therapeutic interventions are available early enough to reduce the downstream morbidity and mortality attributable to hemorrhage, shock and coagulopathy. Due to the time sensitive nature of the treatment of hemorrhage, the ideal resuscitation intervention would entail use of a blood product containing all essential hemostatic components, closest to time of injury, where prevention or reversal of the devastating downstream consequences of shock and coagulopathy can occur. This proposal will characterized the efficacy of whole blood resuscitation initiated in the prehospital setting to patients in hemorrhagic shock which represents this ideal intervention post-injury. These results will have great potential to dramatically change the way trauma resuscitation occurs today.

DETAILED DESCRIPTION:
Traumatic injury represents an incredible health care burden in the United States and worldwide. Hemorrhage is estimated to be responsible for over 40% of all trauma-related deaths. Ongoing traumatic blood loss is complicated by the well-known 'lethal triad' of coagulopathy, hypothermia and acidosis which results in further unbridled hemorrhage. Uncontrolled bleeding, resultant shock and organ dysfunction remain the leading causes of early in-hospital mortality. Despite advances in trauma resuscitation, a paucity of therapeutic interventions are available early enough to reduce the downstream morbidity and mortality attributable to hemorrhage, shock and coagulopathy.

In-hospital resuscitation of traumatic hemorrhage has changed over the past decade. The underlying principle of current resuscitation practice focuses on preventing or reversing the effects of coagulopathy with the early use of a balanced component transfusion strategy (1:1:1 - plasma: packed red blood cells: platelets). This reconstituted strategy has also been coined 'whole blood-like' resuscitation despite being inferior compositionally to whole blood. The use of whole blood was historically the gold standard for treating hemorrhagic shock during World War I and II, prior to sweeping changes in blood banking practice. Whole blood use continues today and is thought to provide the bleeding patient the identical components they are losing with maximal resuscitative and hemostatic effects.

Recent military experiences continue to show the benefits of fresh whole blood resuscitation demonstrating significant survival and hemostatic advantages. Whole blood has also been postulated to improve microcirculatory hemodynamics, reduce the 'storage lesion' effect and minimize donor exposure risks. A recent civilian study has also demonstrated benefit using modified whole blood after arrival to the hospital where appropriate blood typing and cross matching was performed prior to transfusion. Due to the time sensitive nature of the treatment of hemorrhage, the ideal resuscitation intervention would entail use of a blood product containing all essential hemostatic components, closest to time of injury, where prevention or reversal of the devastating downstream consequences of shock and coagulopathy can occur.

Initiation of whole blood resuscitation in the prehospital setting and continued through the in-hospital phase of treatment to patients in hemorrhagic shock represents this ideal intervention post-injury. Essential to the prehospital initiation of whole blood resuscitation in the civilian population is need for it to be transfused without the need for blood typing or cross matching. Of similar importance is the need for cold storage and recycling of any unused whole blood product, allowing maximal utility of this precious resource.

Based upon the belief that early whole blood resuscitation represents the most efficacious hemostatic resuscitation product for the management of hemorrhage, the University of Pittsburgh is currently utilizing cold stored, low titer, platelet replete-leukocyte reduced, group O whole blood (LTLR-WB) for urgent release in the emergency department, without the need for blood typing or cross matching, for patients in hemorrhagic shock. The hypothesis is that the initiation of LTLR-WB resuscitation in the prehospital setting with continuation through the in-hospital acute resuscitation phase of care will significantly reduce the morbidity and mortality attributable to hemorrhagic shock post-injury as compared to standard prehospital and in-hospital resuscitation practice. Thus, a large pragmatic clinical trial is needed to definitively establish the efficacy and safety of whole blood resuscitation initiated in the prehospital setting. Only a high quality clinical trial will provide the essential evidence to justify and provide the impetus for the use of this precious blood banking resource early post-injury. Because of the challenges associated with execution of these types of large trials particularly in the prehospital setting, it is essential to establish feasibility of this approach in a pilot study and provide experience to inform a definitive large, multicenter whole blood trial. The University of Pittsburgh has a track record of prehospital interventional trials post-injury and the clinical research infrastructure to successfully execute the following this trial.

ELIGIBILITY:
Inclusion Criteria:

Injured patients being transport via an air medical service with hypotension (SBP =/< 90mmHg with tachycardia >108 OR SBP=/<70 without the tachycardia requirement)

Exclusion Criteria:

Age < 18 or > 89 years

Isolated fall from standing injury mechanism

Brain matter exposed or penetrating brain injury (GSW)

CPR > 5 mins with out ROSC

Isolated burns without evidence of traumatic injury

Isolated Drowning or Hanging

No Intravenous or Intraosseous access

Known prisoner or known pregnancy

Referral Hospital Admission

Wearing No PPOWER bracelet

Objection to study voiced by subject or family at scene

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Sperry, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lorence JM, Donohue JK, Iyanna N, Guyette FX, Gimbel E, Brown JB, Daley BJ, Eastridge BJ, Miller RS, Nirula R, Harbrecht BG, Claridge JA, Phelan HA, Vercruysse G, O'Keeffe T, Joseph B, Neal MD, Sperry JL. Characterization of adverse events in injured patients at risk of hemorrhagic shock: a secondary analysis of three harmonized prehospital randomized clinical trials. Trauma Surg Acute Care Open. 2024 Jun 25;9(1):e001465. doi: 10.1136/tsaco-2024-001465. eCollection 2024. PMID 38933603
- [Derived] Guyette FX, Zenati M, Triulzi DJ, Yazer MH, Skroczky H, Early BJ, Adams PW, Brown JB, Alarcon L, Neal MD, Forsythe RM, Zuckerbraun BS, Peitzman AB, Billiar TR, Sperry JL. Prehospital low titer group O whole blood is feasible and safe: Results of a prospective randomized pilot trial. J Trauma Acute Care Surg. 2022 May 1;92(5):839-847. doi: 10.1097/TA.0000000000003551. Epub 2022 Jan 25. PMID 35081595

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LTLR-WB | Standard Care
Started | 40 | 46
Completed | 40 | 46
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LTLR-WB | Standard Care | Total
Number analyzed (Participants) | 40 | 46 | 86
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 46 [27 to 64] | 51 [36 to 62] | 48.5 [33 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 31 | 54
  Male | 17 | 15 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 34 | 43 | 77
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 40 | 46 | 86

OUTCOME MEASURES:

1. Primary Outcome: 28 Day All Cause Mortality
Description: 28 day all cause mortality
Time Frame: 28 days from admission
Measure: Count of Participants; unit: Participants
Arm/Group | LTLR-WB | Standard Care
Number analyzed (Participants) | 40 | 46
Participants | 10 | 12
Statistical Analysis 1: Comparison: LTLR-WB vs Standard Care; Test type: Superiority; p = 0.91, Chi-squared

2. Secondary Outcome: Incidence of Multiple Organ Failure
Description: multiple organ failure using the Denver post-injury MOF score which is a summed score and when the score is 4 or greater from 4 organ system scores, MOF is designated; 4 organ systems (pulmonary [0-3], renal [0-3], hepatic [0-3], cardiovascular [0-3])
Time Frame: 28 days from admission
Measure: Count of Participants; unit: Participants
Arm/Group | LTLR-WB | Standard Care
Number analyzed (Participants) | 40 | 46
Participants | 4 | 9
Statistical Analysis 1: Comparison: LTLR-WB vs Standard Care; Test type: Superiority; p = 0.23, Chi-squared

3. Secondary Outcome: 24 Hour Mortality
Description: 24 hour mortality
Time Frame: 24 hours from admission
Measure: Count of Participants; unit: Participants
Arm/Group | LTLR-WB | Standard Care
Number analyzed (Participants) | 40 | 46
Participants | 6 | 8
Statistical Analysis 1: Comparison: LTLR-WB vs Standard Care; Test type: Superiority; p = 0.76, Chi-squared

ADVERSE EVENTS:
Time Frame: During Hospital admission up to 28 days
Arm/Group | LTLR-WB | Standard Care
All-Cause Mortality (participants affected / at risk) | 10/40 | 12/46
Serious Adverse Events (participants affected / at risk) | 7/40 | 11/46
Other Adverse Events (participants affected / at risk) | 0/40 | 1/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LTLR-WB (N=40) | Standard Care (N=46)
stroke (Nervous system disorders) | 1 (1) | 3 (3)
ARDS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
DVT (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
gastrointestinal bleed (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LTLR-WB (N=40) | Standard Care (N=46)
hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-04): https://cdn.clinicaltrials.gov/large-docs/06/NCT03477006/Prot_SAP_000.pdf